CLINICAL TRIAL: NCT01164735
Title: Topoisomerase 2-Alpha (TOPO2A) Genomic Alterations and Immunohistochemical Expression as Well as Chromosome 17 Polysomy in Advanced or Recurrent Endometrial Carcinoma Treated With Anthracycline-Based Therapy
Brief Title: Biomarkers in Tumor Tissue Samples From Patients With Stage III, Stage IV, or Recurrent Endometrial Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-8013; NCI-2011-02245 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000681556; GOG-8013; GOG-8013 (Other: Gynecologic Oncology Group); GOG-8013 (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Uterine Corpus Carcinoma; Stage III Uterine Corpus Cancer; Stage IV Uterine Corpus Cancer

GROUPS / COHORTS (1):
- Correlative studies: Archived tumor tissue samples are analyzed for topoisomerase 2-alpha gene alteration and expression and chromosome 17 polysomy by FISH and IHC. Clinical information associated with each endometrial carcinoma sample (e.g., age, race/ethnicity, cell type, histologic grade, disease stage, and regimen type) is also collected.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research study is studying biomarkers in tissue samples from patients with stage III, stage IV, or recurrent endometrial cancer. Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the frequency of topoisomerase 2-alpha (TOPO2A) gene copy number alterations (including deletions, gains, and amplification), immunohistochemical expression, and chromosome 17 polysomy in tumor tissue samples from patients with advanced or recurrent endometrial carcinoma treated with anthracycline-based therapy on Gynecologic Oncology Group (GOG)-0177.

II. To assess the relationship between TOPO2A gene copy number alterations, TOPO2A protein expression, chromosome 17 polysomy, and human epidermal growth factor receptor 2 (HER2) status in tumor tissue samples from these patients.

III. To assess the association between TOPO2A status (TOPO2A gene copy number alterations and TOPO2A protein expression), or chromosome 17 polysomy and clinical covariates (e.g., age, race/ethnicity, cell type, histologic grade, disease stage, regimen type).

IV. To assess the association between TOPO2A status or chromosome 17 polysomy with measures of clinical outcome including response, progression-free survival, and overall survival of patients treated with this regimen.

V. To evaluate the potential identification of cut points for TOPO2A protein expression with potential prognostic value in patients treated with this regimen.

OUTLINE:

Archived tumor tissue samples are analyzed for topoisomerase 2-alpha gene alteration and expression and chromosome 17 polysomy by fluorescent in situ hybridization (FISH) and immunohistochemistry (IHC). Clinical information associated with each endometrial carcinoma sample (e.g., age, race/ethnicity, cell type, histologic grade, disease stage, and regimen type) is also collected.

ELIGIBILITY:
Inclusion Criteria:

* Chemotherapy-naïve women with histologically documented measurable Stage III, Stage IV or recurrent endometrial carcinoma with known HER2 status who participated in Gynecologic Oncology Group (GOG)-0177 are eligible
* Patients must have given permission for their archival formalin-fixed, paraffin-embedded primary, metastatic or recurrent tumor to be submitted and used for GOG-0177, and at least one to three unstained slides must be available for FISH analysis of TOPO2A and CEP17 and immunohistochemical staining for TOPO2A

Exclusion Criteria:

* Women who were not eligible or evaluable on GOG-0177
* Patients who do not have at least one unstained slide archival formalin-fixed, paraffin-embedded primary, metastatic or recurrent tumor available for fluorescence in situ hybridization (FISH) analysis of TOPO2A and CEP17 or immunohistochemical expression of TOPO2A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | From enrollment on GOG-0177 to death (regardless of cause) or to the date of last contact for women who were alive, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate and plot the unadjusted survival and progression-free survival time distributions by TOPO2A expression and amplification status.

SECONDARY OUTCOMES:
Clinical response (complete or partial response) | Up to 5 years
  Logistic regression modeling will be used to explore the relationship between clinical response to treatment and both TOPO2A expression and amplification.
Progression-free survival | From enrollment on GOG-0177 to disease progression or death, or to the date of last contact for women who were still alive with no evidence of disease progression, assessed up to 5 years
  The Kaplan-Meier method will be used to estimate and plot the unadjusted survival and progression-free survival time distributions by TOPO2A expression and amplification status.

CONTACTS AND LOCATIONS:
Overall Officials: Tatyana Grushko, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Grushko TA, Filiaci VL, Montag AG, Apushkin M, Gomez MJ, Monovich L, Ramirez NC, Schwab C, Kesterson JP, Seward SM, Method MW, Olopade OI, Fleming GF, Birrer MJ. Effects of Slide Storage on Detection of Molecular Markers by IHC and FISH in Endometrial Cancer Tissues From a Clinical Trial: An NRG Oncology/GOG Pilot Study. Appl Immunohistochem Mol Morphol. 2022 Jan 1;30(1):27-35. doi: 10.1097/PAI.0000000000000949. PMID 34224438